CLINICAL TRIAL: NCT05244213
Title: Neoadjuvant Sintilimab Plus Chemotherapy in EGFR-mutant Stage II-IIIB NSCLC: A Single-arm, Open-label Prospective Study
Brief Title: Neoadjuvant Immunotherapy in EGFR-mutant Localized NSCLC
Acronym: NEOTIDE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTONG2104
Record Dates: First submitted 2022-02-08; First posted 2022-02-17 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Non-small Cell Lung Cancer; EGFR Activating Mutation
Keywords: Neoadjuvant immunotherapy; Non-small cell lung cancer; EGFR mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sintilimab; Carboplatin; Taxes

STUDY DESIGN:
Intervention Model Description: A Simon two-stage design was applied. Primary endpoint for this study was MPR. The unacceptable response rate for MPR was less than 10% and desirable response rate was 30%. The error rate for alpha was set as 0.05 and 0.1 for beta. The Optimal assay was chosen and at least 35 patients should be enrolled to meet adequate statical power. 18 patients would be enrolled in stage I and at least 2 patient achieved MPR were required to proceed stage II enrollment. Overall, if 6 achieved MPR out of 35 patients, the study would be determined as positive.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab plus chemo (Experimental): 3 cycles of neoadjuvant Sintilimab (200mg every 3 weeks) with nab-paclitaxel and carboplatin (nab-paclitaxel 260 mg/m2, d1 and carboplatin AUC 5, d1 every 3 weeks) will be administered before surgery, followed by optional adjuvant treatment including EGFR-TKIs for up to 1 year or till disease progression or unacceptable toxicity.
  Interventions: Biological: Sintilimab; Drug: Carboplatin; Drug: Nab paclitaxel

INTERVENTIONS:
Biological: Sintilimab — 200mg Q3W
Drug: Carboplatin — AUC 5, d1 every 3 weeks
Drug: Nab paclitaxel — 260 mg/m2, d1 every 3 weeks

SUMMARY:
Phase II, single-arm, open-label single center study that assess clinical feasibility and safety of 3 cycles neoadjuvant Sintilimab plus chemotherapy in EGFR-mutant stage IIB-IIIB NSCLC (excluding N3) followed by optional adjuvant treatment upon investigators' decisions.

DETAILED DESCRIPTION:
35 eligible patients will be enrolled and 3 cycles of Sintilimab 200mg + doublet platinum-based chemotherapy will be administered. Dynamic blood samples before, during or after neoadjuvant treatment will be obtained for exploratory analysis. Patients who showed inferior response to neoadjuvant treatment leading to unresectable disease will be scheduled for local radiation or other potential subsequent treatment regarding multidisciplinary discussion. After completion of local treatment (surgery or radiation), patients will be provided with optional adjuvant treatment including EGFR-TKI upon investigators' consideration. Patients will be followed with 5 years after surgery. The primary objective of the study is major pathological response (MPR) defined as no more than 10% residual tumor found in primary lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age :18 Years to 75 Years;
2. ECOG physical score 0-1 points; expected survival time ≥ 3 months;
3. Pathologically confirmed diagnosis with Stage II-IIIB(N2) NSCLC which harbored sensitive and rare EGFR alteration. Suspected N2 disease should be confirmed by either mediastinoscopy or EBUS. N1 disease could be determined through PET/CT but biopsy of primary lung cancer is needed;
4. At least one measurable target lesion according to the RECIST 1.1 standard;
5. The main organ function meets the following criteria: 1) blood routine: absolute value of neutrophils ≥ 1.5 × 109 / L, platelets ≥ 75 × 109 / L, hemoglobin ≥ 80 g / L; 2) blood biochemistry: total bilirubin ≤ 1.5 times the upper limit of normal value, aspartate aminotransferase and alanine aminotransferase ≤ 2.5 times the upper limit of normal value (if liver metastasis, ≤ upper limit of normal value 5 times), serum creatinine ≤ 1.5 times the upper limit of normal;
6. Subjects voluntarily joined the study and signed informed consent, with good compliance to follow-up.

Exclusion Criteria:

1. Stage I and stage IV NSCLC;
2. Large panel NGS indicated ALK fusion or any other driver mutations;
3. Histologically confirmed small cell lung cancer (including lung cancer mixed with small cell lung cancer and non-small cell lung cancer);
4. Patients who have previously used any other anti-tumor drugs or radiotherapy;
5. A history of active bleeding within the 6 months before enrollment, or receiving thrombolysis or anticoagulant therapy, or the investigator believes that there is a clear tendency to gastrointestinal bleeding (such as esophageal varices with bleeding risk, local activity) Ulcer lesions, etc.) or active hemoptysis;
6. Patients with any underlying disease that investigators consider it may affect patient's prognosis including sever cardiovascular, pulmonary disease or serious infections;
7. Clinically obvious gastrointestinal abnormalities, which may affect the intake, transport or absorption of drugs (such as inability to swallow, chronic diarrhea, intestinal obstruction, etc.), or patients with total gastrectomy;
8. Pregnant or lactating women; those who have fertility are unwilling or unable to take effective contraceptive measures;
9. Patients with low compliance or willingness to take the drugs and surveillance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-06-04 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Major Pathological Response (MPR) | MPR will be assessed within 2 weeks after surgery
  Percentage of Participants with Major Pathologic Response. MPR was defined as percentage of tumor cells within tumor bed less than 10% for primary lung lesions.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Tumor response will be evaluated within 3-4 weeks after last dose of neoadjuvant treatment
  ORR is the number of participants with a Complete Response (CR) and Partial Response (PR) divided by the total number of randomized participants per arm, then multiplied by 100. Response is based on the Response Evaluation Criteria In Solid Tumors (RECIST 1.1) criteria. Complete Response (CR) was defined as the disappearance of all target lesions. Partial Response (PR) was defined as at least a 30% decrease in sum of longest diameter of target lesions compared to baseline or the complete disappearance of target lesions, with persistence of 1 or more nontarget lesion(s) and no new lesions.
Pathological Complete Response (pCR) | pCR will be assessed within 2 weeks after surgery
  Evaluation of the pathological complete response: The pathological complete response is defined as the absence of residual tumor in both lung and lymph nodes after neoadjuvant treatment.
Progression-free Survival (PFS) | From date of initiation of neoadjuvant treatment till the date of first documented disease progression or death, whichever came first, assessed up to 36 months.
  The period after initiation of neoadjuvant treatment when no disease progression can be detected.
Overall Survival (OS) | From date of initiation of neoadjuvant treatment till the date of all-cause death, assessed up to 60 months.
  The period after initiation of neoadjuvant treatment when no all-cause death can be detected.
Adverse Events (AEs) | From date of initiation of neoadjuvant treatment till treatment discontinuation, assessed up to 14 weeks.
  Incidence of all grade AE which has been confirmed to be correlated with neoadjuvant treatment

CONTACTS AND LOCATIONS:
Overall Officials: Wen-zhao Zhong, PhD, Principal Investigator — Guangdong Lung Cancer Institute, Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Lung Cancer Institute, Guangdong Provincial People's Hospital, Guangdong Academy of Medical Sciences, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
After the primary data including translational analysis has been published, IPD of detailed clinical information and comics data could be available from principle investigator upon reasonable request.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: After the primary data including translational analysis has been published, IPD of detailed clinical information and comics data could be available. Approximate 48 months after initiation of enrollment.
Access Criteria: IPD could be accessed from principle investigator upon reasonable request.

REFERENCES:
- [Background] Shu CA, Gainor JF, Awad MM, Chiuzan C, Grigg CM, Pabani A, Garofano RF, Stoopler MB, Cheng SK, White A, Lanuti M, D'Ovidio F, Bacchetta M, Sonett JR, Saqi A, Rizvi NA. Neoadjuvant atezolizumab and chemotherapy in patients with resectable non-small-cell lung cancer: an open-label, multicentre, single-arm, phase 2 trial. Lancet Oncol. 2020 Jun;21(6):786-795. doi: 10.1016/S1470-2045(20)30140-6. Epub 2020 May 7. PMID 32386568
- [Background] Provencio M, Nadal E, Insa A, Garcia-Campelo MR, Casal-Rubio J, Domine M, Majem M, Rodriguez-Abreu D, Martinez-Marti A, De Castro Carpeno J, Cobo M, Lopez Vivanco G, Del Barco E, Bernabe Caro R, Vinolas N, Barneto Aranda I, Viteri S, Pereira E, Royuela A, Casarrubios M, Salas Anton C, Parra ER, Wistuba I, Calvo V, Laza-Briviesca R, Romero A, Massuti B, Cruz-Bermudez A. Neoadjuvant chemotherapy and nivolumab in resectable non-small-cell lung cancer (NADIM): an open-label, multicentre, single-arm, phase 2 trial. Lancet Oncol. 2020 Nov;21(11):1413-1422. doi: 10.1016/S1470-2045(20)30453-8. Epub 2020 Sep 24. PMID 32979984
- [Background] Forde PM, Chaft JE, Smith KN, Anagnostou V, Cottrell TR, Hellmann MD, Zahurak M, Yang SC, Jones DR, Broderick S, Battafarano RJ, Velez MJ, Rekhtman N, Olah Z, Naidoo J, Marrone KA, Verde F, Guo H, Zhang J, Caushi JX, Chan HY, Sidhom JW, Scharpf RB, White J, Gabrielson E, Wang H, Rosner GL, Rusch V, Wolchok JD, Merghoub T, Taube JM, Velculescu VE, Topalian SL, Brahmer JR, Pardoll DM. Neoadjuvant PD-1 Blockade in Resectable Lung Cancer. N Engl J Med. 2018 May 24;378(21):1976-1986. doi: 10.1056/NEJMoa1716078. Epub 2018 Apr 16. PMID 29658848
- [Background] Reck M, Mok TSK, Nishio M, Jotte RM, Cappuzzo F, Orlandi F, Stroyakovskiy D, Nogami N, Rodriguez-Abreu D, Moro-Sibilot D, Thomas CA, Barlesi F, Finley G, Lee A, Coleman S, Deng Y, Kowanetz M, Shankar G, Lin W, Socinski MA; IMpower150 Study Group. Atezolizumab plus bevacizumab and chemotherapy in non-small-cell lung cancer (IMpower150): key subgroup analyses of patients with EGFR mutations or baseline liver metastases in a randomised, open-label phase 3 trial. Lancet Respir Med. 2019 May;7(5):387-401. doi: 10.1016/S2213-2600(19)30084-0. Epub 2019 Mar 25. PMID 30922878
- [Background] Zhang C, Chen HF, Yan S, Wu L, Yan LX, Yan XL, Yue DS, Xu CW, Zheng M, Li JS, Liu SY, Yang LL, Jiang BY, Ou QX, Qiu ZB, Shao Y, Wu YL, Zhong WZ. Induction immune-checkpoint inhibitors for resectable oncogene-mutant NSCLC: A multicenter pooled analysis. NPJ Precis Oncol. 2022 Sep 19;6(1):66. doi: 10.1038/s41698-022-00301-8. PMID 36123526